CLINICAL TRIAL: NCT01186419
Title: A Phase 2, 24 Week, Randomized, Open Label, Multi-Center Study to Assess the Safety, Tolerability, and Pharmacodynamics of FBS0701 in the Treatment of Chronic Iron Overload Requiring Chelation Therapy, With a 72 Week Dosing Extension
Brief Title: Safety and Pharmacodynamic Study of an Oral Iron Chelator Given for 6 Months to Patients With Iron Overload
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPD602-201; 2010-019645-25 (EudraCT Number); FBS0701-CTP-04 (Other: Ferrokin)
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Results first posted 2015-06-03 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Transfusional Iron Overload; Beta-thalassemia
Keywords: Beta-thalassemia; Sickle cell anemia; Transfusional iron overload; Iron overload; Iron chelation
MeSH Terms: conditions — beta-Thalassemia; Anemia, Sickle Cell; Iron Overload | interventions — 4,5-dihydro-2-(2-hydroxy-3-(3,6,9-trioxadecyloxy)phenyl)-4-methyl-4-thiazolecarboxylic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPD602 (16mg) (Experimental)
  Interventions: Drug: SPD602 (FBS0701, SSP-004184)
- SPD602 (32mg) (Experimental)
  Interventions: Drug: SPD602 (FBS0701, SSP-004184)

INTERVENTIONS:
Drug: SPD602 (FBS0701, SSP-004184) — Oral FBS0701 taken one time daily for up to 96 weeks.

SUMMARY:
The purpose of this research study is to evaluate the safety of two doses of FBS0701, a new oral iron chelator, and its effectiveness in clearing iron from the liver. FBS0701 is a medication taken by mouth that causes the body to get rid of iron. Iron chelators are used in patients with β-thalassemia and other forms of anemia who experience iron overload - iron increases in the body as a result of regularly required blood transfusions. Patients who qualify will be randomized to receive one of two doses of FBS0701 for up to 24 weeks (6 months) with a total study duration of up to 33 weeks. These patients will be eligible to participate in a dosing extension for up to 72 weeks. The maximum duration of dosing will be up to 96 weeks. The safety of patients will be monitored frequently during the study by physical exams, ECGs, and blood tests. To assess the amount of iron in the liver and heart, each patient must undergo 6 MRI scans during the study. Patients will not need to stay in the hospital for this study but will need to visit the outpatient clinic up to 28 times over the 96 week period. Patients currently taking an iron chelator will be required to stop for a total of up to 26 weeks. The results of this study will help to determine if FBS0701 may be effective as an iron chelator.

ELIGIBILITY:
Inclusion Criteria:

* Transfusional iron overload due to: hereditary anemias such as sickle cell disease, β-thalassemia and Diamond-Blackfan anemia; acquired anemias such as Myelodysplastic Syndrome and other forms of bone marrow failure. Patients must also be transfusion-dependent and require chronic treatment with deferoxamine, deferasirox, and/or deferiprone.
* Willing to discontinue all existing iron chelation therapies throughout study period.
* Serum ferritin greater than 500 ng/mL at Screening.
* Baseline liver iron concentration and cardiac MRI T2* per protocol requirements.
* Mean of the previous three pre-transfusion hemoglobin concentrations greater than or equal to 7.5 g/dL.
* Agrees to use an approved method of contraception throughout study period.

Exclusion Criteria:

* As a result of medical review, physical examination or Screening investigations, the Principal Investigator considers the patient unfit for the study.
* Non-elective hospitalization within the 30 days prior to Baseline testing. (Patients with sickle cell anemia who are admitted to the hospital for management of sickle crisis pain whose uncomplicated hospital course was four days or less and who, 14 days prior to Baseline testing, have returned to their previous health status are acceptable.)
* Evidence of clinically relevant oral, cardiovascular, gastrointestinal, hepatic, renal, endocrine, pulmonary, neurologic, psychiatric, immunologic, bone marrow or skin disorder as determined by the Investigator.
* Evidence of significant renal insufficiency; possible examples include: serum creatinine above the upper limit of normal, proteinuria greater than 2 gm per day or calculated creatinine clearance of less than 60 mL/minute.
* Cardiac left ventricular ejection fraction outside of protocol requirements.
* Known sensitivity to magnesium stearate, croscarmellose sodium or FBS0701.
* Platelet count below 100,000/µL and/or absolute neutrophil count less than 1500/mm3 at Screening and <50% at Baseline testing by MRI
* Alkaline phosphatase, AST or ALT outside of protocol requirements.
* Liver Function Tests: ALT >5 times the local upper limit of normal on two occasions in the previous 12 months or ALT at Screening >200 IU/L
* Use of any investigational agent within the 30 days prior to the Baseline testing.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2010-08-13 (Actual); Primary Completion 2013-01-08 (Actual); Study Completion 2013-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (9):
- United States (2):
  - Children's Hospital and Research Center of Oakland, Oakland, California
  - Children's Hospital of Boston, Boston, Massachusetts
- Italy (3):
  - Ospedale Regionale Microcitemie, Cagliari
  - Centro della Microcitemia e delle Anemie Congenite, Genoa
  - Thalassemia Center San Luigi Hospital, Orbassano
- Siriraj Hospital, Mahidol University, Bangkok, Thailand
- Pediatric Hematology, Ege University Hospital, Izmir, Turkey (Türkiye)
- United Kingdom (2):
  - University College London Hospital, London
  - Whittington Hospital, London

REFERENCES:
- [Derived] Padhani ZA, Gangwani MK, Sadaf A, Hasan B, Colan S, Alvi N, Das JK. Calcium channel blockers for preventing cardiomyopathy due to iron overload in people with transfusion-dependent beta thalassaemia. Cochrane Database Syst Rev. 2023 Nov 17;11(11):CD011626. doi: 10.1002/14651858.CD011626.pub3. PMID 37975597
- [Derived] Wood JC, Zhang P, Rienhoff H, Abi-Saab W, Neufeld E. R2 and R2* are equally effective in evaluating chronic response to iron chelation. Am J Hematol. 2014 May;89(5):505-8. doi: 10.1002/ajh.23673. Epub 2014 Mar 3. PMID 24452753
- [Derived] Neufeld EJ, Galanello R, Viprakasit V, Aydinok Y, Piga A, Harmatz P, Forni GL, Shah FT, Grace RF, Porter JB, Wood JC, Peppe J, Jones A, Rienhoff HY Jr. A phase 2 study of the safety, tolerability, and pharmacodynamics of FBS0701, a novel oral iron chelator, in transfusional iron overload. Blood. 2012 Apr 5;119(14):3263-8. doi: 10.1182/blood-2011-10-386268. Epub 2012 Jan 17. PMID 22251482
- [Derived] Rienhoff HY Jr, Viprakasit V, Tay L, Harmatz P, Vichinsky E, Chirnomas D, Kwiatkowski JL, Tapper A, Kramer W, Porter JB, Neufeld EJ. A phase 1 dose-escalation study: safety, tolerability, and pharmacokinetics of FBS0701, a novel oral iron chelator for the treatment of transfusional iron overload. Haematologica. 2011 Apr;96(4):521-5. doi: 10.3324/haematol.2010.034405. Epub 2010 Dec 20. PMID 21173101

RESULTS

PARTICIPANT FLOW:
Groups:
- SPD602 16 mg/kg/Day; SPD602 32 mg/kg/Day: Participants received SPD602 orally once daily for up to 96 weeks. At Week 24, the iron clearing activity of SPD602 was assessed for each participant and the dose may have been adjusted to a higher or lower dose if the clinical response was deemed insufficient or too robust, respectively (maximum dose=60mg/kg/day; minimum dose=8mg/kg/day). Participants not dose adjusted at Week 24 may also have had later dose adjustments to a higher or lower dose.
Period: Overall Study
Arm/Group | SPD602 16 mg/kg/Day | SPD602 32 mg/kg/Day
Started | 24 | 27
Completed | 17 | 18
Not Completed | 7 | 9
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Physician Decision | 0 | 3
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: All subjects who received any amount of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | SPD602 16 mg/kg/Day | SPD602 32 mg/kg/Day | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 24 | 26 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (8.60) | 28.4 (7.11) | 28.5 (7.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Liver Iron Concentration (LIC) at 96 Weeks
Description: LIC was determined by R2 Magnetic Resonance Imaging (MRI).
Time Frame: Baseline and 96 weeks
Population: Full Analysis Set, defined as all subjects in the Safety Set who had at least 1 post-baseline primary efficacy assessment. The Safety Set was defined as all subjects who received any amount of investigational product.
Measure: Mean (Standard Deviation); unit: mg/g
Groups:
- SPD602: Participants received SPD602 orally once daily for up to 96 weeks.
Arm/Group | SPD602
Number analyzed (Participants) | 26
mg/g | -1.75 (4.839)
Statistical Analysis 1: Comparison: SPD602; Test type: Superiority or Other; p = 0.0765, t-test, 2 sided

2. Secondary Outcome: Maximum Plasma Concentration (Cmax) of SPD602
Description: Cmax is a term that refers to the maximum (or peak) concentration that a drug achieves in the body after the drug has been administered.
Time Frame: 92 weeks
Population: Pharmacokinetic (PK) Analysis Set, defined as all subjects in the Safety Set for whom the primary PK data were considered sufficient and interpretable. The Safety Set was defined as all subjects who received any amount of investigational product.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | SPD602
Number analyzed (Participants) | 5
ng/ml | 25702.7 (4448.06)

3. Secondary Outcome: Area Under The Steady-state Plasma Concentration-time Curve (AUC) of SPD602
Description: AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure of how much and how long a drug stays in a body.
Time Frame: 92 weeks
Population: PK Analysis Set, defined as all subjects in the Safety Set for whom the primary PK data were considered sufficient and interpretable. The Safety Set was defined as all subjects who received any amount of investigational product.
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | SPD602
Number analyzed (Participants) | 5
ng*hr/ml | 62998.6 (23094.72)

ADVERSE EVENTS:
Groups:
- SPD602 16 mg/kg/d; SPD602 32 mg/kg/d: Participants received SPD602 orally once daily for up to 96 weeks. At Week 24, the iron clearing activity of SPD602 was assessed for each participant and the dose may have been adjusted to a higher or lower dose if the clinical response was deemed insufficient or too robust, respectively (maximum dose=60mg/kg/day; minimum dose=8mg/kg/day). Participants not dose adjusted at Week 24 may also have had later dose adjustments to a higher or lower dose.
Arm/Group | SPD602 16 mg/kg/d | SPD602 32 mg/kg/d
Serious Adverse Events (participants affected / at risk) | 3/24 | 2/27
Other Adverse Events (participants affected / at risk) | 24/24 | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPD602 16 mg/kg/d (N=24) | SPD602 32 mg/kg/d (N=27)
Sickle cell anemia with crisis (Congenital, familial and genetic disorders) | 1 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPD602 16 mg/kg/d (N=24) | SPD602 32 mg/kg/d (N=27)
Palpitations (Cardiac disorders) | 2 (2) | 3 (4)
Conjunctivitis (Eye disorders) | 2 (2) | 2 (2)
Ocular icterus (Eye disorders) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 5 (7)
Colitis (Gastrointestinal disorders) | 1 (1) | 2 (3)
Constipation (Gastrointestinal disorders) | 1 (2) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 5 (7) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 3 (4)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (2)
Asthenia (General disorders) | 3 (4) | 1 (4)
Fatigue (General disorders) | 2 (2) | 1 (2)
Influenza like illness (General disorders) | 2 (3) | 4 (9)
Pyrexia (General disorders) | 4 (7) | 3 (6)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis (Infections and infestations) | 3 (3) | 3 (3)
Influenza (Infections and infestations) | 2 (5) | 6 (7)
Nasopharyngitis (Infections and infestations) | 5 (5) | 4 (4)
Pharyngitis (Infections and infestations) | 5 (5) | 5 (6)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 2 (3)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 3 (3) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 5 (7) | 7 (13)
Viral infection (Infections and infestations) | 1 (1) | 2 (2)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 3 (3)
Cardiac murmur (Investigations) | 0 (0) | 4 (8)
Gamma-glutamyltransferase increased (Investigations) | 1 (4) | 3 (3)
Transaminases increased (Investigations) | 2 (2) | 5 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (10) | 4 (11)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 8 (24) | 9 (15)
Paraesthesia (Nervous system disorders) | 2 (5) | 4 (5)
Chromaturia (Renal and urinary disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (10) | 4 (7)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Joint sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Cystitis (Infections and infestations) | 2 (2) | 0 (0)
Oral herpes (Infections and infestations) | 2 (2) | 0 (0)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 2 (7) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (9) | 0 (0)

LIMITATIONS AND CAVEATS:
Only data from all subjects (ie, total) are presented because dose adjustments that occurred after Week 24 obviated the meaningful interpretation of data presented by the original 16 and 32 mg/kg/day dose groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.